CLINICAL TRIAL: NCT00003332
Title: Phase I/II Study of Induction Chemotherapy With Gemcitabine and Cisplatin Followed by Combined Chemo-radiation and/or Surgical Resection for Locally Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy Followed by Chemotherapy and Radiation Therapy and/or Surgery in Treating Patients Who Have Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066296; P30CA016087 (NIH); NYU-9703; NCI-G98-1423
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cisplatin; Gemcitabine; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug with radiation therapy and/or surgery may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy, consisting of gemcitabine and cisplatin, followed by chemotherapy and radiation therapy and/or surgery in treating patients who have pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with locally advanced pancreatic cancer after induction therapy with gemcitabine and cisplatin.
* Determine the maximum tolerated dose of gemcitabine and cisplatin chemotherapy combined with radiation therapy in these patients.
* Determine the overall response rates in these patients after this combined modality regimen following induction chemotherapy.
* Determine the resectability rate for locally advanced pancreatic lesions treated with this regimen.
* Determine the time to failure for the entire treatment program.

OUTLINE: This is a dose-escalation study.

Patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Following gemcitabine, patients receive cisplatin IV over 1 hour on days 1, 8, and 15. Course is repeated every 4 weeks. After 2 courses of induction chemotherapy, disease is restaged.

Patients may then receive radiotherapy in addition to chemotherapy. Radiotherapy is given daily for 5 weeks and 3 days. During radiotherapy, cohorts of 3 patients are treated with escalating doses of gemcitabine and cisplatin administered as described above in induction chemotherapy. The maximum tolerated dose (MTD) is defined as the lowest dose at which no more than 2 of 6 or 2 of 3 patients experience dose limiting toxicity. When the MTD has been determined, additional patients accrued into the study receive the dose level immediately below the MTD.

If after 2 courses of induction chemotherapy with gemcitabine and cisplatin the tumor is radiographically considered resectable by operating surgeon, the patient undergoes surgical exploration or laparoscopy for staging and verification of resectability. If the tumor is found to be resectable without evidence of distant disease, the patient undergoes complete surgical resection and radiation plus adjuvant gemcitabine and cisplatin.

Patients are followed every 3 months until death.

PROJECTED ACCRUAL: Approximately 15-36 patients will be accrued for the Phase I portion of this study and there will be 14-25 patients accrued into the Phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed localized adenocarcinoma of the pancreas that is considered unresectable
* Measurable or evaluable disease
* No metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin less than 3.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min

Other:

* No serious concurrent systemic disorder
* No active infection or uncontrolled infection
* Not pregnant
* Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Other:

* At least 1 month since any prior investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-07; Primary Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States